CLINICAL TRIAL: NCT03357497
Title: Very Early Mobilization of Colorectal Surgery Patients - A Randomized Controlled Trial
Brief Title: Very Early Mobilization of Colorectal Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 230961
Record Dates: First submitted 2017-09-25; First posted 2017-11-30 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Care; Colorectal Surgery
Keywords: colorectal surgery, early mobilization, postoperative care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very early mobilization (Experimental): This group will be mobilized in the post-operative unit by a designated physiotherapist. The intervention will be conducted accordingly with the SOMS protocol.
  Interventions: Other: Very early mobilization
- Standard post-operative care (No Intervention): This group will receive standard post-operative care. Mobilization will only take place if the patient request it or to facilitate god post-operative care.

INTERVENTIONS:
Other: Very early mobilization — The patient will be mobilized by a physiotherapist in our postoperative care unit. The intervention uses the SOMS protocol.
  Arms: Very early mobilization

SUMMARY:
Early mobilization is an important part of Enhanced Recovery Programs (ERP)in colorectal surgery. The aim of this randomized controlled trial is to investigate the impact of very early mobilization, starting within 1 hour after surgery, on further mobilization within an existing Enhanced Recovery Program.

DETAILED DESCRIPTION:
Post-operative bed rest and immobility has a negative effect on morbidity and mortality after colorectal surgery.To prevent immobilization early mobilization is a well established part of Enhanced Recovery Programs. This facility uses protocols developed by the ERAS (Enhanced Recovery After Surgery)-society. However not all patients can reach the level physical activity needed to be in compliance with the ERP. This being more frequent in the elderly frail patient. This may contribute to longer hospital stay and increase the risk of complications. The aim of this trial is to investigate if a very early mobilization intervention will lead to a higher lever of physical activity after surgery compared with standard-care.

The aim is to include 150 patients scheduled to undergo colorectal surgery. Patients will receive written and verbal information about the trial before written consent is obtained. The patients will undergo an extended pre-operative assessment during which a baseline for patients physical activity level will be established before surgery. For this purpose the patients will be evaluated by a physiotherapist with the following tools; 6-minutes walk test, Timed up and go-test (TUG), mini modified Functional Independence Measure (mFIM), WHO disability assessment score (WHODAS) and activity measurement with accelerometry for up to 7 days. (Actigraph GT3X device)

The randomization will take place on the day of the surgery and the patients will be assigned to either intervention (very early mobilization) or control group (standard post-operative care). A stratified randomization will be performed to ensure an even spread within three patient categories: Laparoscopic surgery, Open surgery and Rectum amputation. The randomization is performed using concealed allocation where envelopes are prepared externally using a randomization list prepared by a statistician.

After surgery the patients will be transferred to the post-operative care unit where the patients included in the intervention group will be mobilized with the help of a physiotherapist and post-operative unit staff. The intervention will begin as early as 30 minutes after arrival in the post-operative unit. The intervention will follow the Surgical ICU Optimal Mobilization Score (SOMS) which includes four steps of mobilization from movement in bed up to walking. Progress from each step to the next will be conditioned with patient fulfilling criteria for a safe mobilization including stable physiological parameters and adequate pain situation. The patients in the standard care group will not receive the intervention.

All patients will receive information about early mobilization. The patients will not receive information on the timing of the mobilization intervention in an effort to remain blinded to the intervention. The patient in the standard care group will be mobilized accordingly to the ERP protocol, which also includes early mobilization in the surgical ward. Upon transfer from the post-operative unit to the surgical ward all study patients will be again fitted with the activity monitor to measure their physical activity during the post-operative phase.

During hospital stay all study patients will be subject to routine mobilization within the existing ERP protocol. To determine the physical activity level the patient will be wearing the activity monitoring device until discharge from the surgical ward. The study patients will also be evaluated by blinded physiotherapists with mFIM and 6 minutes walk-test. In addition information will be gathered regarding routine documentation on patient mobilization progress to measure adherence to ERP goals.

After four to six weeks the patients are scheduled for a standard post-operative follow-up visit. The study patients will then also meet a blinded physiotherapist that previously was not participating in the intervention who will repeat the following tests: 6 minutes walk-test, WHODAS, TUG. All study patients will also be instructed to wear the activity monitor for additional seven days to again measure their physical activity level. All patients who have undergone the intervention will be scheduled for a semi-structured telephone interview about their perception of the SOMS intervention.

Follow-up questionnaire with WHODAS self-reported questions will be gathered through a telephone interview with the patients three, six and twelve months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 scheduled for colorectal surgery

Exclusion Criteria:

* Unable to understand study information (language,cognitive impairment, etc.)
* Unable to walk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Physical activity level measured with accelerometry | 72 hours
  Comparison between intervention and standard-care group by measurements of physical activity level with an accelerometer that the patient wears during the day. The accelerometer is worn at hip level.

SECONDARY OUTCOMES:
Time out of bed measured with a protocol | 7 days
  Comparison between intervention and standard-care group, analysis of time out of bed and thus compliance to ERP goals using written documentation in the surgical ward.
Minutes in the postoperative ward | one year
  To ascertain if this intervention is cost effective by comparing time in the post-operative unit between intervention and standard care group.
Days in the hospital ward | one year
  To ascertain if this intervention is cost effective by comparing total hospital stay time between intervention and standard care group.
Number of adverse events during the SOMS intervention. | one day
  Frequency of adverse events during the intervention using the SOMS-protocol. Adverse events here are abnormal blood pressure, pulse, oxygen saturation %, respiratory rate, pain, presence of vertigo, presence of nausea and vomiting.
Blood pressure during the SOMS intervention. | one day
  Blood pressure are registered during the intervention.
Pulse during the SOMS intervention. | one day
  Number of heartbeats are registered during the intervention with a device on the patients finger.
Oxygen saturation during the SOMS intervention. | one day
  Oxygen saturation are registered during the intervention with a device on the patients finger.
Pain | one day
  Pain experienced by the patient during the SOMS intervention, rated using a Visual analogue scale 0-100.
Presence of vertigo | one day
  Vertigo experienced by the patient during the SOMS intervention, presence rated as yes/no.
Presence of nausea | one day
  Nausea experienced by the patient during the SOMS intervention, presence rated as yes/no. If patient vomits due to nausea is also rated yes/no.
6 minute Walking test | 6 weeks
  Physical capacity measured with the 6 minute Walking test. The number of meters a patient walks during 6 minutes.
Timed up and Go (TUG) test | 6 weeks
  Test of functional mobility. The patient sits on a chair, rises and walks 3 meters, turns och walks back and sits down on the chair. Time in seconds to perform the test.
Patient perception of the SOMS intervention | 6 weeks
  Semi structured telephone interview with patients in the intervention group about their perception of the intervention.
Severity of post-operative complications | one year
  Monitoring number and frequency of patient complications with review of patient records using Clavien-Dindo complication classification
Self-perceived health and physical function level one year after surgery | one year
  Using the WHODAS questionnaire, self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ahlstrand, M.D. PhD, Principal Investigator — Region Örebro län; Anette Forsberg, PhD, Principal Investigator — Region Örebro län
Locations (1):
- Universitetssjukhuset Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harper CM, Lyles YM. Physiology and complications of bed rest. J Am Geriatr Soc. 1988 Nov;36(11):1047-54. doi: 10.1111/j.1532-5415.1988.tb04375.x. PMID 3049751
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Smart NJ, White P, Allison AS, Ockrim JB, Kennedy RH, Francis NK. Deviation and failure of enhanced recovery after surgery following laparoscopic colorectal surgery: early prediction model. Colorectal Dis. 2012 Oct;14(10):e727-34. doi: 10.1111/j.1463-1318.2012.03096.x. PMID 22594524
- [Background] Castelino T, Fiore JF Jr, Niculiseanu P, Landry T, Augustin B, Feldman LS. The effect of early mobilization protocols on postoperative outcomes following abdominal and thoracic surgery: A systematic review. Surgery. 2016 Apr;159(4):991-1003. doi: 10.1016/j.surg.2015.11.029. Epub 2016 Jan 21. PMID 26804821
- [Background] Shulman MA, Myles PS, Chan MT, McIlroy DR, Wallace S, Ponsford J. Measurement of disability-free survival after surgery. Anesthesiology. 2015 Mar;122(3):524-36. doi: 10.1097/ALN.0000000000000586. PMID 25689757
- [Background] Meyer MJ, Stanislaus AB, Lee J, Waak K, Ryan C, Saxena R, Ball S, Schmidt U, Poon T, Piva S, Walz M, Talmor DS, Blobner M, Latronico N, Eikermann M. Surgical Intensive Care Unit Optimal Mobilisation Score (SOMS) trial: a protocol for an international, multicentre, randomised controlled trial focused on goal-directed early mobilisation of surgical ICU patients. BMJ Open. 2013 Aug 19;3(8):e003262. doi: 10.1136/bmjopen-2013-003262. PMID 23959756
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Keith RA, Granger CV, Hamilton BB, Sherwin FS. The functional independence measure: a new tool for rehabilitation. Adv Clin Rehabil. 1987;1:6-18. No abstract available. PMID 3503663
- [Derived] Thorn RW, Stepniewski J, Hjelmqvist H, Forsberg A, Ahlstrand R, Ljungqvist O. Supervised Immediate Postoperative Mobilization After Elective Colorectal Surgery: A Feasibility Study. World J Surg. 2022 Jan;46(1):34-42. doi: 10.1007/s00268-021-06347-2. Epub 2021 Oct 19. PMID 34668047